CLINICAL TRIAL: NCT00314574
Title: A Phase IIIb Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Xolair in Subjects With Moderate to Severe Persistent Asthma Who Are Inadequately Controlled With High-Dose Inhaled Corticosteroids and Long-Acting Beta-Agonists
Brief Title: A Study of Omalizumab (Xolair) in Subjects With Moderate to Severe Persistent Asthma (EXTRA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q3662g
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Persistent Asthma; EXTRA; Xolair; Difficult Breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Omalizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Xolair (Experimental): The subcutaneous dose of Xolair administered in this study was either a minimum of 0.008 mg/kg/IgE (IU/mL) every 2 weeks or a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks for 48 weeks.
  Participants maintained their high-dose inhaled corticosteroid (minimum of 500 µg of fluticasone dry powder inhaler twice a day or its ex-valve equivalent) and Long-Acting Beta-Agonist dose (either 50 µg salmeterol twice daily or 12 µg formoterol twice daily) throughout the study.
  Participants were permitted to use albuterol as rescue medicine throughout the study.
  Interventions: Drug: omalizumab (Xolair); Drug: corticosteroids; Drug: long-acting beta-agonists
- placebo (Placebo Comparator): The subcutaneous dose of placebo administered in this study was either a minimum of 0.008 mg/kg/IgE (IU/mL) every 2 weeks or a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks for 48 weeks.
  Participants maintained their high-dose inhaled corticosteroid (minimum of 500 µg of fluticasone dry powder inhaler twice a day or its ex-valve equivalent) and Long-Acting Beta-Agonist dose (either 50 µg salmeterol twice daily or 12 µg formoterol twice daily) throughout the study.
  Participants were permitted to use albuterol as rescue medicine throughout the study.
  Interventions: Drug: placebo; Drug: corticosteroids; Drug: long-acting beta-agonists

INTERVENTIONS:
Drug: omalizumab (Xolair) — Omalizumab (Xolair) was administered by subcutaneous (SC) injection every 2 or 4 weeks. Xolair was supplied as a sterile, white, preservative-free, lyophilized powder in single-use vials that were reconstituted with Sterile Water for Injection (SWFI), USP.
  Other Names: Xolair
  Arms: Xolair
Drug: placebo — Placebo was administered by subcutaneous (SC) injection every 2 or 4 weeks. Placebo contained the same ingredients as the lyophilized formulation of Xolair,excluding omalizumab.
  Arms: placebo
Drug: corticosteroids — Minimum dose of 500 µg of fluticasone dry-powder inhaler or its equivalent ex-valve dose twice a day.
Drug: long-acting beta-agonists — 50 µg salmeterol twice daily or 12 µg formoterol twice daily.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study of the efficacy, safety, and tolerability of subcutaneously administered Xolair as add-on therapy for the treatment of subjects aged 12-75 years old diagnosed with moderate to severe asthma who are inadequately controlled with high-dose inhaled corticosteroids (ICS)+ long-acting beta-agonists (LABA) with or without additional controller therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form and an informed assent, if applicable
* Be between the ages of 12 to 75 years
* Have had a history of moderate to severe asthma for at least one year prior to screening
* Have had treatment with a stable regimen of of salmeterol 50 µg twice a day (BID) or formoterol 12 µg BID for at least 8 weeks prior to screening
* Have had treatment with a stable regimen of high-dose inhaled corticosteroids (ICS) for at least 8 weeks prior to screening
* Have inadequately controlled asthma
* Have had at least one asthma exacerbation requiring systemic corticosteroid rescue in the 12 months prior to the screening visit while receiving treatment with high-dose ICS
* Have less than 10 pack-years smoking history
* Have a positive skin test for or a positive, in vitro response to one relevant perennial aeroallergen documented within the 12 months prior to screening
* If a subject has not had a positive skin test or in vitro reactivity in the 12 months prior to screening, the subject must demonstrate a positive response to at least one relevant perennial aeroallergen in a skin or in vitro test prior to randomization
* Female subjects of childbearing potential must use an effective method of contraception from screening through their duration of participation in the study
* For the collection of additional blood samples for future research (optional), provide signed consent and an informed assent, if applicable.

Exclusion Criteria:

* Have had an asthma exacerbation requiring intubation within 12 months prior to screening
* Have active lung disease other than asthma
* Have had an asthma exacerbation requiring treatment with the addition of systemic (oral or intravenous) corticosteroids or an increase in systemic corticosteroids within 30 days prior to screening
* Require chronic immunosuppressive therapy including cyclosporine, methotrexate, etc.
* Have significant medical illness other than asthma
* Have taken methotrexate, gold salts, cyclosporine, or macrolide antibiotics, within 3 months prior to screening
* Have taken other investigational drugs within 30 days prior to screening
* Have been treated with Xolair within the 12 months prior to screening
* Have a history of drug or alcohol abuse that, in the judgment of the investigator, may put the subject at risk for being unable to participate fully in the study for the duration of the study
* Have elevated serum IgE levels for reasons other than allergy
* Are pregnant or lactating

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2005-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Rosen, M.D., Ph.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Szefler SJ, Jerschow E, Yoo B, Janampally P, Pazwash H, Holweg CTJ, Hudes G. Response to Omalizumab in Black and White Patients with Allergic Asthma. J Allergy Clin Immunol Pract. 2021 Nov;9(11):4021-4028. doi: 10.1016/j.jaip.2021.07.013. Epub 2021 Jul 22. PMID 34303017
- [Derived] Chen M, Choo E, Yoo B, Raut P, Haselkorn T, Pazwash H, Holweg CTJ, Hudes G. No difference in omalizumab efficacy in patients with asthma by number of asthma-related and allergic comorbidities. Ann Allergy Asthma Immunol. 2021 Jun;126(6):666-673. doi: 10.1016/j.anai.2021.01.015. Epub 2021 Jan 17. PMID 33465457
- [Derived] Busse WW, Szefler SJ, Haselkorn T, Iqbal A, Ortiz B, Lanier BQ, Chipps BE. Possible Protective Effect of Omalizumab on Lung Function Decline in Patients Experiencing Asthma Exacerbations. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1201-1211. doi: 10.1016/j.jaip.2020.10.027. Epub 2020 Oct 24. PMID 33223095
- [Derived] Chen M, Shepard K 2nd, Yang M, Raut P, Pazwash H, Holweg CTJ, Choo E. Overlap of allergic, eosinophilic and type 2 inflammatory subtypes in moderate-to-severe asthma. Clin Exp Allergy. 2021 Apr;51(4):546-555. doi: 10.1111/cea.13790. Epub 2021 Jan 7. PMID 33217063
- [Derived] Busse WW, Humbert M, Haselkorn T, Ortiz B, Trzaskoma BL, Stephenson P, Garcia Conde L, Kianifard F, Holgate ST. Effect of omalizumab on lung function and eosinophil levels in adolescents with moderate-to-severe allergic asthma. Ann Allergy Asthma Immunol. 2020 Feb;124(2):190-196. doi: 10.1016/j.anai.2019.11.016. Epub 2019 Nov 22. PMID 31760132
- [Derived] Hanania NA, Wenzel S, Rosen K, Hsieh HJ, Mosesova S, Choy DF, Lal P, Arron JR, Harris JM, Busse W. Exploring the effects of omalizumab in allergic asthma: an analysis of biomarkers in the EXTRA study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):804-11. doi: 10.1164/rccm.201208-1414OC. PMID 23471469
- [Derived] Hanania NA, Alpan O, Hamilos DL, Condemi JJ, Reyes-Rivera I, Zhu J, Rosen KE, Eisner MD, Wong DA, Busse W. Omalizumab in severe allergic asthma inadequately controlled with standard therapy: a randomized trial. Ann Intern Med. 2011 May 3;154(9):573-82. doi: 10.7326/0003-4819-154-9-201105030-00002. PMID 21536936

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo subcutaneous dose minimum of 0.008 mg/kg/IgE (IU/mL) every 2 weeks or a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks for 48 weeks.
  Participants maintained their high-dose inhaled corticosteroid (minimum of 500 µg of fluticasone dry powder inhaler twice a day or its ex-valve equivalent) and Long-Acting Beta-Agonist dose (either 50 µg salmeterol twice daily or 12 µg formoterol twice daily) throughout the study.
  Participants were permitted to use albuterol as rescue medicine throughout the study.
- Xolair: Omalizumab (Xolair) subcutaneous dose minimum of 0.008 mg/kg/IgE (IU/mL) every 2 weeks or a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks for 48 weeks.
  Participants maintained their high-dose inhaled corticosteroid (minimum of 500 µg of fluticasone dry powder inhaler twice a day or its ex-valve equivalent) and Long-Acting Beta-Agonist dose (either 50 µg salmeterol twice daily or 12 µg formoterol twice daily) throughout the study.
  Participants were permitted to use albuterol as rescue medicine throughout the study.
Period: Overall Study
Arm/Group | Placebo | Xolair
Started | 423 | 427
Received at Least One Dose of Study Drug | 421 | 427
Safety Population | 420 (1 patient in the placebo arm received Xolair and was added to the Xolair arm for Safety analyses.) | 428
Completed | 329 | 344
Not Completed | 94 | 83
Not completed — Death | 3 | 0
Not completed — Adverse Event | 11 | 16
Not completed — Lost to Follow-up | 19 | 25
Not completed — Withdrawal by Subject | 33 | 22
Not completed — Physician Decision | 22 | 15
Not completed — Pregnancy | 6 | 4
Not completed — Data unknown at database lock | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Xolair | Total
Number analyzed (Participants) | 421 | 427 | 848
Age, Categorical [Count of Participants; unit: Participants] — All baseline measures were based on all randomized subjects who received at least one dose of study drug (the modified ITT population). The modified ITT population included 848 subjects (427 subjects in the Xolair group and 421 subjects in the placebo group).
  Participants
    <=18 years | 16 | 23 | 39
    Between 18 and 65 years | 376 | 379 | 755
    >=65 years | 29 | 25 | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.9) | 43.7 (14.3) | 44.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 262 | 557
  Male | 126 | 165 | 291

OUTCOME MEASURES:

1. Primary Outcome: Rate of Asthma Exacerbations Over the 48 Week Treatment Period
Description: A protocol-defined asthma exacerbation was defined as worsening of asthma symptoms requiring treatment with systemic corticosteroids for 3 or more days; for patients receiving long-term oral corticosteroids, an exacerbation was a 20 mg or more increase in average daily dose of oral prednisone (or a similar dose of another systemic corticosteroid). The rate of protocol-defined asthma exacerbations, normalized by subject-time at risk and computed over the 48 week treatment period in each treatment group.
Time Frame: 48 weeks
Population: Modified Intent-to-Treat population included all randomized patients who received at least 1 dose of study drug (Xolair or placebo).
Measure: Number; unit: exacerbation/patient-week
Arm/Group | Placebo | Xolair
Number analyzed (Participants) | 421 | 427
exacerbation/patient-week | 0.88 [0.6139 to 0.9212] | 0.66 [0.6139 to 0.9212]

2. Secondary Outcome: Change From Baseline in Total Asthma Symptom Scores
Description: Change from baseline to week 48 in Total Asthma Symptom Score (TASS), which included a nocturnal asthma score (0 to 4 scale), morning asthma symptoms (yes or no), and a daytime asthma symptom score (0 to 4 scale, total score range 0 to 9, higher TASS scores represent worse symptoms; breathlessness, tightness in chest, wheezing and cough. Score achieved by week 48 minus baseline.
Time Frame: Baseline and Week 48
Population: Modified Intent-to-Treat population included all randomized patients who received at least 1 dose of study drug. Ten patients were missing baseline values and were excluded from the analyses. The Last Observation Carried Forward was used to impute missing values at week 48 for patients who discontinued the study early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Xolair
Number analyzed (Participants) | 417 | 421
score on a scale | -1.36 (1.87) [-0.49 to -0.01] | -1.61 (1.85) [-0.49 to -0.01]

3. Secondary Outcome: Change From Baseline in the Number of Puffs Per Day of Beta Agonist Rescue Medication
Description: Change from baseline to week 48 in mean puffs per day of albuterol. Puffs per day was achieved by week 48 minus baseline.
Time Frame: Baseline and Week 48
Population: Modified Intent-to-Treat population included all randomized patients who received at least 1 dose of study drug (Xolair or placebo). Five patients were missing baseline values and were excluded from the analyses. The Last Observation Carried Forward was used to impute missing values at week 48 for patients who discontinued the study early.
Measure: Mean (Standard Deviation); unit: puffs per day
Arm/Group | Placebo | Xolair
Number analyzed (Participants) | 417 | 426
puffs per day | -1.35 (2.69) | -1.57 (2.58)

4. Secondary Outcome: Change From Baseline in Overall Asthma-related Quality of Life
Description: Change from baseline to week 48 in overall asthma-specific health-related quality of life, as measured by the standardized version of the Asthma Quality of Life Questionnaire (AQLQ[S]) score. The AQLQ(S) consists of 4 domains (activity limitations, symptoms, emotional function, and environmental stimuli), with a total of 32 items; the overall score is the mean of these 32 items on a scale of 1 to 7 (1 = severe impairment, 7 = no impairment). Overall outcome achieved by mean visit minus baseline.
Time Frame: Baseline and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Xolair
Number analyzed (Participants) | 418 | 425
score on a scale | 0.96 (1.26) [0.07 to 0.39] | 1.16 (1.22) [0.07 to 0.39]

5. Secondary Outcome: Number of Participants Assessed for Frequency and Severity of Treatment-emergent Adverse Events
Description: This outcome is represented in the adverse event section of the database.
Time Frame: Week 48
Population: Safety Population: The safety-evaluable population comprised 848 patients (428 Xolair group and 420 placebo group). Patients in the safety-evaluable population were analyzed according to the actual treatment received. One subject was assigned to receive placebo but inadvertently received at least one dose of xolair during the study.
Measure: Number; unit: participants
Arm/Group | Placebo | Xolair
Number analyzed (Participants) | 420 | 428
participants | 420 | 428

ADVERSE EVENTS:
Time Frame: 48 Weeks
Description: The safety-evaluable population, used for all safety analyses, included all randomized subjects who received at least one study drug. Subjects were analyzed according to the actual treatment received. One subject was assigned to receive placebo but inadvertently received at least one dose of xolair during the study.
Arm/Group | Placebo | Xolair
Serious Adverse Events (participants affected / at risk) | 44/420 | 40/428
Other Adverse Events (participants affected / at risk) | 339/420 | 329/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=420) | Xolair (N=428)
iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0
atrial fibrillation (Cardiac disorders) | 2 | 0
coronary artery disease (Cardiac disorders) | 0 | 1
arrhythmia (Cardiac disorders) | 1 | 0
cardiac arrest (Cardiac disorders) | 1 | 0
pancreatitis (Gastrointestinal disorders) | 0 | 1
pancreatitis acute (Gastrointestinal disorders) | 0 | 1
hiatus hernia (Gastrointestinal disorders) | 1 | 0
irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
intestinal obstruction (Gastrointestinal disorders) | 1 | 0
chest pain (General disorders) | 3 | 2
bile duct stenosis (Hepatobiliary disorders) | 0 | 1
anaphylactic reaction (Immune system disorders) | 1 | 0
diverticulitis (Infections and infestations) | 1 | 1
appendicitis (Infections and infestations) | 0 | 1
gastroenteritis (Infections and infestations) | 0 | 1
pneumonia (Infections and infestations) | 2 | 1
lobar pneumonia (Infections and infestations) | 0 | 1
gastroenteritis viral (Infections and infestations) | 1 | 1
meningitis viral (Infections and infestations) | 0 | 1
respiratory tract infection (Infections and infestations) | 1 | 0
wound infection (Infections and infestations) | 0 | 1
influenza (Infections and infestations) | 2 | 0
chronic sinusitis (Infections and infestations) | 1 | 0
sinusitis (Infections and infestations) | 0 | 1
kidney infection (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 1 | 0
cellulitis (Infections and infestations) | 1 | 0
vaginal abscess (Infections and infestations) | 1 | 0
fall (Injury, poisoning and procedural complications) | 0 | 1
open wound (Injury, poisoning and procedural complications) | 0 | 1
open fracture (Injury, poisoning and procedural complications) | 1 | 0
urinary bladder rupture (Injury, poisoning and procedural complications) | 1 | 0
facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
rib fracture (Injury, poisoning and procedural complications) | 0 | 1
forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 1
headache (Nervous system disorders) | 0 | 1
amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
bipolar disorder (Psychiatric disorders) | 0 | 1
bipolar I disorder (Psychiatric disorders) | 0 | 1
depression (Psychiatric disorders) | 1 | 0
renal failure (Renal and urinary disorders) | 1 | 0
nephrolithiasis (Renal and urinary disorders) | 0 | 1
uterine enlargement (Reproductive system and breast disorders) | 1 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 17
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 1 | 0
deep vein thrombosis (Vascular disorders) | 1 | 1
hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=420) | Xolair (N=428)
sinusitis (Infections and infestations) | 79 | 81
bronchitis (Infections and infestations) | 60 | 66
nasopharyngitis (Infections and infestations) | 38 | 36
acute sinusitis (Infections and infestations) | 19 | 23
influenza (Infections and infestations) | 17 | 22
urinary tract infection (Infections and infestations) | 25 | 20
upper respiratory infection (Infections and infestations) | 93 | 96
back pain (Musculoskeletal and connective tissue disorders) | 23 | 15
headache (Nervous system disorders) | 34 | 41
cough (Respiratory, thoracic and mediastinal disorders) | 29 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."